CLINICAL TRIAL: NCT00813735
Title: Eszopiclone Co-Administered With Escitalopram for Insomnia in Elderly Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lehigh Center for Clinical Research (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESRCO66
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Insomnia
Keywords: Insomnia; Major Depression; Geriatric
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major | interventions — Eszopiclone; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eszopiclone (Experimental): Drug: Eszopiclone 2mg, Drug: Escitalopram 10mg or 20mg
  Interventions: Drug: Eszopiclone; Drug: Escitalopram
- Placebo (Placebo Comparator): Drug: Placebo, Drug: Escitalopram 10mg or 20mg
  Interventions: Drug: Placebo; Drug: Escitalopram

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 2mg daily at bedtime
  Other Names: Escitalopram 10mg or 20mg daily in the AM
  Arms: Eszopiclone
Drug: Placebo — Placebo daily at bedtime
  Other Names: Escitalopram 10mg or 20mg daily in the AM
  Arms: Placebo
Drug: Escitalopram — Escitalopram 10mg or 20mg

SUMMARY:
Research has established the incidence of insomnia increases with age and the possible causes contributing to sleep problems in the elderly are still being explored and debated. Older adults use a disproportionately large share of sleep aids with non-prescription sleep aid use having increased over the past decade. This study is a double blind safety and effectiveness trial examining the response of eszopiclone co-administered with escitalopram for the treatment of insomnia symptoms in geriatric depressed adults with insomnia symptoms.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, parallel-group study. There are two groups of subjects with Major Depressive Disorder and insomnia symptoms randomized to treatment either with eszopicone 2mg or placebo daily at bedtime for 14 weeks beginning at visit 2. Also, all subjects receive open label treatment with escitalopram 10 or 20mg daily in the morning. Safety and efficacy is evaluated as well as rating scales and patient sleep diaries.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDD, HAMD score 20 or greater at screening and baseline, total sleep time less than 6 hours at screening and baseline, ISI 15 or greater at screening and baseline

Exclusion Criteria:

* May not use any other psychoactive drugs/psychotropics during study, may not have any type of dementia, may not have any significant/unstable medical problems, no nightshift work permitted, no current seizure disorders/head injuries

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in total sleep time from baseline to final visit | from baseline to final visit

SECONDARY OUTCOMES:
change in sleep latency from baseline to final visit | from baseline to final visit
Change in HAMD from baseline to final visit | from baseline to final visit
Change in ISI from baseline to final visit | baseline to final visit
Change in CGI-S, CGI-I from baseline to final visit | baseline to final visit
labs (CBC,urinalysis,TSH,Chemprofile,drugscreen),height | visit 1
vitals: BP,pulse,temperature,weight,assess AE's/SAE's | every visit

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Gross, Principal Investigator — Lehigh Center for Clinical Research
Locations (1):
- Lehigh Center for Clinical Research, Allentown, Pennsylvania, United States